CLINICAL TRIAL: NCT02378649
Title: A Randomized, Placebo Controlled, Single Center Clinical Trial for Evaluation of Efficacy and Safety of Sildenafil Administration in the Cardiac ICU Following Mitral Valve Surgery in Patients With Pulmonary Hypertension
Brief Title: PDEI Following Mitral Valve Surgery in Patients With Pulmonary Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dr. Robert Klempfner Heart Rehabilitation Institute (Other Government)
Responsible Party: Sponsor-Investigator, Dr. Robert Klempfner Heart Rehabilitation Institute, Dr. Ferstenfeld Ido, Sheba Medical Center
Organization: Sheba Medical Center (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1839-14-SMC
Record Dates: First submitted 2015-02-05; First posted 2015-03-04 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Pulmonary Hypertension; Mitral Valve Surgery
Keywords: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Sildenafil (Experimental): PDEI or placebo will be administered in the surgical ICU 4-6 hours after arriving from the Operative Room. The initial Dose will be 20mg X 3 NG and can be increase to 40mg X 3, it will be administered PO if the patient extubated.
  PDEI or placebo will continue up to 8 days or discharge.
  Interventions: Drug: Sildenafil
- Placebo (Placebo Comparator): PDEI or placebo will be administered in the surgical ICU 4-6 hours after arriving from the Operative Room. The initial Dose will be 20mg X 3 NG and can be increase to 40mg X 3, it will be administered PO if the patient extubated.
  PDEI or placebo will continue up to 8 days or discharge.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sildenafil — Sildenafil administration in the cardiac ICU following Mitral Valve Surgery concomitant with best practice usual care
  Other Names: Revatio \ Viagra
  Arms: Sildenafil
Drug: Placebo — Placebo comparator concomitant with best practice usual care
  Arms: Placebo

SUMMARY:
A randomized, placebo controlled, single center clinical trial for evaluation of efficacy and safety of Sildenafil administration in the cardiac ICU following Mitral Valve (MV) Surgery in patients with pre-operative Significant Pulmonary Hypertension.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 22
2. Undergoing mitral valve surgery (either repair or replacement) with or without coronary revascularization, aortic valve replacement (AVR) or repair; or tricuspid valve surgery.
3. Pre-operative pulmonary arterial systolic pressure >50 mm Hg as determined by resting echocardiography and post-operative sPAP > 45 mmHg as obtained from invasive hemodynamics measurements.
4. Willing and able to give written informed consent prior to the procedure

Exclusion Criteria:

1. Hypersensitivity to study drug
2. Women of child-bearing potential
3. Expected need to administer nitrates that are clinically indicated peri-operatively
4. Post-operative hypotension (systolic blood pressure (BP) <80) or evidence of shock (postoperative evidence of any kinds of shock)
5. Cardiac or systemic amyloidosis
6. Active malignancy other than BCC (basal cell carcinoma)
7. Stable kidney dysfunction with Creatine clearence (CrCl) <30 mL/min during the screening period or hepatic failure other than mild
8. Significant anemia (hemoglobin <8 mg/dl) preoperative.
9. Known drug or alcohol dependence or any other factors which will interfere with the study conduct or interpretation of the results or in the opinion of the investigator are not suitable to participate;
10. Any illness other than cardiac which might reduce life expectancy to less than 1 year from screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
To evaluate if sildenafil results in greater reduction in average mean pulmonary artery pressure (mPAP) compared to placebo. (Percent change in mPAP pressure at 48 hours as compared to the immediate post operative averages.) | 48 hours
  Percent change in mPAP pressure at 48 hours as compared to the immediate post operative averages. Pulmonary pressures will be obtained through invasive hemodynamic measurements

SECONDARY OUTCOMES:
Time on mechanical ventilation | 96 hours
Total surgical intensive care time | participants will be followed for the duration of ICU stay, an expected average of 4 days
  Duration of Surgical ICU stay
Change in functional capacity post operation (Change in NYHA functional class (optional 6MWT pre-discharge) | participants will be followed for the duration of hospital stay, an expected average of 6 days
  Change in NYHA functional class (optional 6 minute walk test [6MWT] pre-discharge)
Study treatment related serious adverse events | participants will be followed for the duration of hospital stay, an expected average of 6 days
  Absence of serious adverse events related to study drug (shock, organ hypoperfusion, significant arrythmia and any other major event as defined by GCP guidelines) during hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiac Surgical Department, Leviev Heart Center, Ramat Gan, Tel Hashomer, Israel